CLINICAL TRIAL: NCT03501017
Title: The Effect of Physical Activity Performed Under the Guidance of Nurse to the Individuals With Moderate Risk of Cardiovascular Disease on Decreasing Risk Level: Randomized Controlled Study
Brief Title: The Effect of Physical Activity on Decreasing Risk Level
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 00001
Record Dates: First submitted 2018-04-02; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: CVD Risk; Physical Activity; Nurse's Role; Risk Reduction
MeSH Terms: conditions — Motor Activity; Risk Reduction Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The 12-week physical activity program was implemented under the guidance of nurse, in outdoors with the group, 5 days a week with warm up and cooling down for 10 minutes and normal walking tempo at a moderate pace for 30-45 minutes (3-6 km/hour).
  Interventions: Other: physical activity program
- Control Group (Active Comparator): As routine practice, a brochure provided from the Public Health Directorate on protection from CVD was delivered to the individuals in the control group.
  Interventions: Other: Routine Practice

INTERVENTIONS:
Other: physical activity program — The 12-week physical activity program was implemented under the guidance of nurse, in outdoors with the group, 5 days a week with warm up and cooling down for 10 minutes and normal walking tempo at a moderate pace for 30-45 minutes (3-6 km/hour).
  Application of WHO Smoking Cessation Algorithm: After fagerström test was applied, the modified smoking cessation algorithm of WHO was applied to the individuals and those who decided to quit smoking were referred to smoking cessation outpatient clinics.
  Arms: Intervention group
Other: Routine Practice — As routine practice, a brochure provided from the Public Health Directorate on protection from CVD was delivered to the individuals in the control group.
  Arms: Control Group

SUMMARY:
Objective: The aim of the first part of this study with two stages is to determine prevalence of CVD risk and the associated variables in individuals aged 40-65 years registered in a Family Health Center (FHC) in city center of Antalya; the aim of the second one is to evaluate the effect of intervention to increase physical activity in individuals with moderate risk of CVD on decreasing the risk level.

Methods: Stage 1 and Stage 2 were conducted as cross-sectional and Randomized Controlled Experimental Trial, respectively.

In the first stage the CVD risk level was calculated using the HeartScore. In the second stage, 11 individuals with moderate CVD risk (2-<5%) found in the intervention group participated into a 12-week physical activity program (a moderate walk outdoor, with group 5 days in a week, each lasting for 40 minutes) guided by nurse. CVD brochure and physical activity guide was distributed to 11 individuals in control group within the scope of routine practice of FHCs.

DETAILED DESCRIPTION:
The purpose of this study is to determine Cardiovascular Disease (CVD) risk level in 40-65 year-old individuals coming to a FHC and to evaluate the effect of increasing the physical activity and interventions about the changeable risk factors on reducing the risk level in individuals with moderate CVD risk.

Hypothesis; the 12-week group walking activity about changing CVD risk factors reduces the risk level more in intervention group compared to the control group (H1).

It provides blood pressure control in the intervention group. It reduces cholesterol. It helps reducing the weight, BMI, and waist circumference values. This study was conducted in two stages. Stage 1: In order to determine the high risk prevalence of CVD, it was carried out in Akdeniz FHC located in Konyaalti Central District of Antalya between April and September 2016.

Stage 2: In order to evaluate the effect of the interventions for the changeable risk factors (HeartScore 2-<5%) in individuals with moderate level of CVD risk, the study was conducted as a Randomized Controlled Experimental Trial between October-December 2016 in April 23 Park located near to FHC in the same region. There is a hiking trail around this park. This trail is 860-meter long, covered with rubber, and suitable for walking. In addition, there are two fields for exercise on apparatus in the east and west side of the park.

Stage 1 Population and Sample The population of the study consisted of 2390 individuals aged between 40 and 65 years registered in the Akdeniz FHC. In the study, the sample size was calculated by considering the CVD moderate risk prevalence (27.4%) obtained by Ünal et al. in their study conducted with individuals living in Balcova region via the formula used in the cases of known population and the minimum sample size for this study was determined as 27012. However, 327 individuals were voluntary to participate in the study between the dates when the study was conducted and their risk levels were calculated by using HeartScore® program.

Stage 2 Population and Sample Seventy two individuals who were found to have moderate risk as a result of the first stage of the study constituted the population of this stage. 22 people met the inclusion criteria of the study. When the sample size power was evaluated with Power and Sample Size Calculation program for determining the difference between two dependent numerical variables with the power of 80% and the error margin of 0.05 in Randomized Controlled Trials (RCT), it was determined that minimum 9 people is sufficient for each group.

Preliminary preparation The content of the study was explained to the individuals meeting the inclusion criteria of the study in detail.

Current CVD risks of the individuals determined as the intervention group were re-measured before the physical activity program and it was emphasized that their current risk can be reduced after the 12-week program.

In order to encourage individuals to participate in physical activity programs, materials such as pedometer, hats, and t-shirts were distributed before starting the program.

The feature of pedometer distributed to the individuals to keep time and distance of the conducted activity was used. The necessary technical settings for the pedometer were made by the researcher daily and weekly.

Healthy Beverage Distribution

•Individuals were asked to come with empty stomach and water was distributed before the walk so that they could meet their fluid needs. They were advised to drink at least 2.5-3 liters of water per day. In addition, in order to encourage the individuals to healthy diet, "ayran" (a drink made with yoghurt and water), milk and mineral water were regularly distributed in certain periods every day.

Intervention: 12-Week Physical Activity Program Physical activity program was administered to all individuals in the experimental group whose risk was found as 2-<5% by evaluating their all risk factors using HeartScore® program. In this direction, International Physical Activity Questionnaire (IPAQ Short Form) was first applied to the individuals in order to determine again their physical activity levels. Individuals determined to be inactive and minimally active according to this measure were included in the physical activity program recommended by the Ministry of Health and International Guidelines as a nonpharmacological tool in primary prevention of CVD.

Duration of moderate intensity physical activity or aerobic exercise which can reduce total and cardiovascular mortality are 2.5 - 5 hours a week; as the total period of the weekly physical activity prolonged, the observed benefits increased as well. For this reason, physical activity program was completed in such a way to complete minimum 150 minutes per week. It was explained that the time individuals need to walk per week should be minimum 150 minutes. However, some individuals increased this time up to 200-250 minutes per week according to their availability and willingness statuses.

With the pedometer distributed to the individuals, step, distance, pace and the calories burned were recorded and these records were taken daily with the table prepared specific for the individuals. The aim here was to increase their motivation by showing them the developments in their physical activity levels. In addition, thanks to the record feature of pedometer, the extra steps taken by individuals who wanted to continue to walk could be recorded, the steps taken by the individuals who could not continue to walk due to personal reasons (being sick, hospital appointment, etc.) and walked individually on that day were also recorded.

In order to regularly determine the weight lost by the individuals and to increase their motivations, Mondays in each week were determined as "Scale Day" and weight and waist circumference values were measured and the obtained values were recorded.

Application of WHO Smoking Cessation Algorithm After fagerström test was applied, the modified smoking cessation algorithm of World Health Organization (WHO) was applied to the individuals and those who decided to quit smoking were referred to smoking cessation outpatient clinics. For the individuals who decided to quit smoking, appointments were made from the smoking cessation outpatient clinic located in Cancer Early Detection, Screening and Education Center which provides free services.

Routine Practice for Control Group As routine practice, a brochure provided from the Public Health Directorate on protection from CVD was delivered to the individuals in the control group.

As the posttest to the individuals after applying the above-planned interventions; HeartScore® risk level assessment, implementation of IPAQ questionnaire, BMI, weight and waist circumference measurements were performed.

ELIGIBILITY:
Inclusion Criteria:

* Being aged between 40 and 65 years,
* Not having a problem that could prevent walking activity,
* Being voluntary to participate in the study.

Exclusion Criteria:

* Having a known and diagnosed CVD, being diagnosed with diabetes (they are evaluated to have a high risk in the European Guidelines on Cardiovascular Disease Prevention and treatment is recommended),
* Having walking disabled,
* Not being voluntary to participate in the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2016-06-20 (Actual); Primary Completion 2016-10-25 (Actual); Study Completion 2016-12-20 (Actual)

PRIMARY OUTCOMES:
Change in CVD risk level | 12 week
  "HeartScore® program" was used to determine the CVD risk level in the first stage of the study. In the second part, the risk level was evaluated using HeartScore program for the second time.
  HeartScore® is a primary prevention tool that provides risk measurement for people who have not had any cardiovascular disease.
  According to the SCORE score calculated in the European Guidelines on Cardiovascular Disease Prevention in Clinical Practice, individuals are divided into 4 risk categories. Accordingly, if SCORE score is;
  * ≥%10, very high risk category,
  * Between ≥%5- <%10, high risk category
  * Between ≥%2- <5, moderate risk category,
  * <%1, then they are in the low risk category.

SECONDARY OUTCOMES:
Change in Opinions and Experiences about Physical Activity | 12 week
  Participants' thoughts and experiences related to physical activity were assessed with a semi-structured interview form. Each participant was interviewed once. The duration of the interview continued to the point where no new information or opinion was obtained.
Change in Physical activity level | 12 week
  Physical activity level was measured by using Short Form of International Physical Activity Questionnaire (IPAQ).
  Short form (7 questions); provides information about the time spent on waking, moderate-intensity and vigorous-intensity activities, and the time spent on sitting. IPAQ classifies individuals categorically as "inactive", "minimally active", and "very active".

CONTACTS AND LOCATIONS:
Overall Officials: Sebahat Gözüm, Prof, Principal Investigator — Akdeniz University

IPD SHARING:
Plan to Share IPD: No